CLINICAL TRIAL: NCT06047899
Title: Influence of the Dietary Supplement Luteolin for Two Weeks on Memory in Healthy Subjects
Brief Title: Influence of Luteolin for Two Weeks on Memory in Healthy Subjects
Acronym: LuMus2-2023
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dominique de Quervain, MD (Other)
Responsible Party: Sponsor-Investigator, Prof. Dominique de Quervain, MD, Director Division of Cognitive Neuroscience, University of Basel
Organization: University of Basel (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2023-01628
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Memory
MeSH Terms: interventions — Luteolin

STUDY DESIGN:
Intervention Model Description: randomized double-blind placebo-controlled cross-over counter-balanced
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): In the intervention phase we will administer 500 mg luteolin (2x250 mg capsules, e.g. every morning and evening) per day formulated for oral administration for 14.5 days.
  Interventions: Dietary Supplement: Luteolin
- Placebo (Placebo Comparator): Placebo control intervention consists of identical looking placebo capsules containing mannitol formulated for oral administration to be taken twice daily (e.g. every morning and evening) for 14.5 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Luteolin — Luteolin extracted from Chrysanthemum Ramat 98% HPLC by Scyherb® food grade certified according to Safe Quality Foods (SQF) - Level 3 Comprehensive Food Safety and Quality Management System Certification by the Safe Quality Food Institute (SQFI).
  Arms: Intervention
Other: Placebo — mannitol formulated for oral administration (capsules)
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn about the effect of the dietary supplement luteolin in healthy people. The main question it aims to answer is: Does luteolin have an influence on memory functions?

Participants will go trough two treatment phases. In one phase they will take 250mg luteolin twice daily for two weeks. In the other phase they will take a placebo twice daily for two weeks. A placebo is a look-alike substance that contains no active drug.

At the start and end of teach treatment phase, participants will undergo different memory testing exercises in our research facility.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* male or female
* able to give written informed consent as documented by signature
* Aged: 18 to 40 years
* normotensive (BP 90/60mmHg to 140/90mmHg)
* BMI ≤ 30 kg/m2

Exclusion Criteria:

* bodyweight <50 kg
* pregnant or lactating women
* intention to become pregnant during the course of the study
* known or suspected non-compliance, drug or alcohol abuse
* MADRS-S total score > 12 or MADRS-S item 9 >1
* inability to follow the procedures of the study, e.g. due to language problems, psychological disorders
* participation in another study with investigational drug within the 30 days preceding and during the present study
* participation in one of our previous studies using the same memory tests in the past 2 years or participation in our first luteolin study in 2020
* enrolment of the investigator, his/her family members, employees and other dependent persons

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2023-11-28 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
Visual Memory Test | short delay (5 minutes), long delay (14 days): to assess differences between these time points
  Performance in a visual memory test (Rey-Osterrieth complex figure test (Rey 1941) and (Osterrieth 1944)). As parallel version we will use the modified complex Taylor figure test (Hubley 2002).
  Participants will have to copy the complex figure. After a short delay of 5 minutes, they will be asked to redraw the figure from memory. A long-delayed recall test will be administered 2 weeks after the learning phase.
  Performance is calculated by scoring for accuracy and relative position of the 18 units in the whole of the design. Maximal score is 36 points.

SECONDARY OUTCOMES:
Verbal Memory Task | immediate recall, short delay (10 minutes), long delay (14 days): to assess differences between these time points
  Verbal memory task (de Quervain, Roozendaal et al. 2000). A parallel version will be used for the second study phase.
  Subjects are given explicit instructions to learn 60 unrelated German nouns for immediate and delayed recall. For all free-recall tests (immediate recall, short delay and long delay), subjects will be asked to write down all the words they remember. The number of correctly recalled words (hits) will be the relevant output.
  Delayed recall of all 60 words will be tested about 10 min (short delay) and 2 weeks (long delay) after presentation.
Working Memory Test | after each treatment phase (duration two weeks)
  Working memory will be assessed with the digit span task backward, a subtest of the "Wechsler Intelligenztest für Erwachsene" (von Aster 2006). A parallel version will be used for each visit. Each correct reproduction of a sequence of numbers is scored with one point.
Mood State (MDBF) | after each treatment phase (duration two weeks)
  Mood state will be assessed with the self-rating instrument MDBF (Steyer 1997) consisting of 12 items to be rated in a 5 scale mode. The total score is calculated by summing the answers in each of the 3 dimensions good/bad mood, alertness/sleepiness, rest /restlessness with 4 items in each dimension. We will use a parallel version for each visit.
Depressive Symptoms | after each treatment phase (duration two weeks)
  Depressive symptoms will be assessed with the self-rating questionnaire MADRS-S (Cunningham 2011) (Schmidtke 1988). This scale consists of 9 items assessing participants' mood, feelings of unease, sleep, appetite, ability to concentrate, initiative, emotional involvement, pessimism and zest for life. Each item is scored between 0 and 3. The total score is calculated by summing the answers of the nine items, ranging between 0 and 27 (higher scores indicate increased impairment).
Anxiety | after each treatment phase (duration two weeks)
  Anxiety will be measured with the self-rating instrument STAI-G form X1 (state) (Laux 1981).This instrument consists of 20 items scored between 1-4. The total score is calculated by summing the answers, ranging between 20 and 80.
Visual Analog Scales Quality of Sleep | after each treatment phase (duration two weeks)
  Subjective sleep quality is assessed using a visual analogue scale (VAS) in relation to the past two weeks. Respondents specify their level of agreement to the statement by indicating a position along a continuous line (10 cm) between the two end-points: better sleep quality respectively than normal or worse. The score ranges between -5 and + 5.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique de Quervain, Prof, Study Chair — University of Basel; Christiane Gerhards, MD, Principal Investigator — University of Basel
Locations (1):
- University of Basel, Division of Cognitive Neuroscience, Basel, Canton of Basel-City, Switzerland